CLINICAL TRIAL: NCT06036121
Title: A Phase 1a/b Study of ADRX-0706 in Subjects With Select Advanced Solid Tumors
Brief Title: A Study of ADRX-0706 in Select Advanced Solid Tumors
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Adcentrx Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ADRX-0706-001
Record Dates: First submitted 2023-09-06; First posted 2023-09-13 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Solid Tumors; Triple Negative Breast Cancer (TNBC); Urothelial Cancer; Cervical Cancer
Keywords: urothelial cancer; triple negative breast cancer; cervical cancer; ADC
MeSH Terms: conditions — Triple Negative Breast Neoplasms; Uterine Cervical Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Phase 1a Dose Escalation (Experimental): Increasing doses of ADRX-0706 will be administered to identify the maximum tolerated dose (MTD) and the recommended dose to be used in the Phase 1b part.
  Interventions: Drug: ADRX-0706
- Phase 1b Dose Expansion (Experimental): ADRX-0706 will be initially administered to patients at the dose recommended from the Phase 1a part in 3 disease-specific cohorts: urothelial cancer, triple negative breast cancer, and cervical cancer.
  Interventions: Drug: ADRX-0706

INTERVENTIONS:
Drug: ADRX-0706 — Antibody drug conjugate targeting Nectin-4

SUMMARY:
The primary purpose of this study is to assess the safety, tolerability, and pharmacokinetics, and to identify the optimal dose of ADRX-0706 in patients with select advanced solid tumors.

DETAILED DESCRIPTION:
This is a 2 part study. The Phase 1a will consist of a dose escalation of ADRX-0706 to evaluate initial safety and tolerability in patients with select advanced solid tumors, and to identify the recommended dose to be used in the Phase 1b. The Phase 1b will further evaluate the safety and tolerability, as well as preliminary efficacy, and identify the optimal dose of ADRX-0706 in patients with urothelial cancer, triple negative breast cancer, and cervical cancer.

ELIGIBILITY:
Inclusion Criteria:

* Phase 1a Dose Escalation: Subjects with histologically confirmed select advanced solid tumors, including urothelial carcinoma (UC), head and neck squamous cell carcinoma (HNSCC), breast cancer, cervical cancer, ovarian cancer, non-small cell lung cancer (NSCLC), and pancreatic cancer. Subjects must have received at least one prior systemic regimen and have no other therapy available known to provide meaningful clinical benefit in the opinion of the investigator.
* Phase 1b Dose Expansion: Subjects with urothelial cancer, triple negative breast cancer or cervical cancer with disease progression after at least one prior systemic regimen and no standard treatment options available and considered appropriate in the opinion of the investigator, unless subject refuses standard therapy.
* Measurable disease according to RECIST version 1.1
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Adequate hematologic, liver, and renal function

Exclusion Criteria:

* Active and uncontrolled central nervous system metastases
* Significant cardiovascular disease
* History of another malignancy other than the one for which the subject is being treated on this study within 3 years
* Receipt of any anticancer or investigational therapy within 5 elimination half-lives or 14 days (whichever is less)
* Any P-gp inducers/inhibitors or strong CYP3A inhibitors received within 14 days prior to the first dose of study drug
* Receiving systemic antimicrobial treatment for active infection; routine antimicrobial prophylaxis is permitted

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2023-09-26 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events | Until study completion (estimated 3 years)

SECONDARY OUTCOMES:
Measurement of maximum plasma concentration (Cmax) of ADRX-0706 | Until study completion (estimated 3 years)
  Measured from pharmacokinetic (PK) blood samples
Measurement of trough concentration (Ctrough) of ADRX-0706 | Until study completion (estimated 3 years)
  Measured from PK blood samples
Measurement of area under the serum concentration-time curve (AUC) of ADRX-0706 | Until study completion (estimated 3 years)
  Measured from PK blood samples
Measurement of terminal half-life (t1/2) of ADRX-0706 | Until study completion (estimated 3 years)
  Measured from PK blood samples
Measurement of systemic clearance (CL) of ADRX-0706 | Until study completion (estimated 3 years)
  Measured from PK blood samples
Measurement of volume of distribution at steady state (Vss) of ADRX-0706 | Until study completion (estimated 3 years)
  Measured from PK blood samples
Incidence of anti-drug antibodies (ADA) | Until study completion (estimated 3 years)
  Measured from ADA blood samples
Measurement of objective response rate (ORR) per RECIST 1.1 | Until study completion (estimated 3 years)
  Percentage of subjects achieving complete response (CR) or partial response (PR)
Measurement of duration of response (DOR) | Until study completion (estimated 3 years)
  Time from first response until first evidence of disease progression (PD) or death from any cause
Measurement of disease control rate (DCR) | Until study completion (estimated 3 years)
  Percentage of subjects achieving CR, PR or stable disease (SD)
Measurement of progression free survival (PFS) | Until study completion (estimated 3 years)
  Time from the start of study drug until first evidence of PD or death from any cause
Measurement of overall survival (OS) | Until study completion (estimated 3 years)
  Time from the start of study drug until death from any cause

CONTACTS AND LOCATIONS:
Locations (21):
- United States (13):
  - USC Norris Comprehensive Cancer Center, Los Angeles, California
  - UCLA, Los Angeles, California
  - Comprehensive Hematology Oncology, St. Petersburg, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Cancer, Detroit, Michigan
  - START Midwest, Grand Rapids, Michigan
  - The Ohio State University Wexner Medical Center, Hilliard, Ohio
  - Stephenson Cancer Center, Oklahoma City, Oklahoma
  - Sarah Cannon Cancer Network, Nashville, Tennessee
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - START San Antonio, San Antonio, Texas
  - START Mountain Region, West Valley City, Utah
- China (8):
  - Beijing University Third Hospital, Beijing
  - Fujian Cancer Hospital, Fujian
  - Sun Yat-sen University Cancer Center, Guangzhou
  - Hunan Cancer hospital, Hunan
  - Shandong Cancer Hospital, Jinan
  - Shanghai East Hospital, Shanghai
  - Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan
  - Wuhan Union Hospital, Wuhan

IPD SHARING:
Plan to Share IPD: No